CLINICAL TRIAL: NCT01238536
Title: Multicenter Randomized Controlled Trial of Epidural Steroid Injections for Spinal Stenosis in Persons 50 and Older
Brief Title: Lumbar Epidural Steroid Injections for Spinal Stenosis Multicenter Randomized, Controlled Trial (LESS Trial)
Acronym: LESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); University of California, San Francisco (Other); Henry Ford Hospital (Other); Harvard Pilgrim Health Care (Other); Harvard Vanguard Medical Associates (Other); University of Colorado, Denver (Other); Mayo Clinic (Other); Stanford University (Other); Massachusetts General Hospital (Other); Virginia Spine Research Institute (Unknown); Oregon Health and Science University (Other); Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janna Friedly, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39023D; R01HS019222-01 (AHRQ)
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Spinal Stenosis; Low Back Pain
Keywords: Epidural Steroid Injection; Low Back Pain; Spinal Stenosis; Elderly
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain | interventions — Anesthetics, Local; Triamcinolone Acetonide; Methylprednisolone Acetate; Betamethasone; Dexamethasone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural Steroid injection (Experimental): Epidural steroid injectate will be 2cc of .25 - 1% lidocaine followed by 1-3 cc of 40 mg/cc Kenalog (i.e. 40-120 mg Kenalog) or an equivalent steroid medication (depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg) in an opaque syringe.
  Intervention: Epidural steroid with local anesthetic injection
  2cc of .25 - 1% lidocaine and glucocorticoid (Kenalog 40-120 mg, depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg)
  Interventions: Procedure: Epidural steroid with local anesthetic injection; Drug: Epidural steroid injection
- Epidural local anesthetic injection (Active Comparator): Intervention: Epidural injectate will be 2cc of .25-1% lidocaine followed by 1-3cc of 1% lidocaine in an opaque syringe.
  Interventions: Procedure: Epidural local anesthetic injection; Drug: Epidural local anesthetic injection

INTERVENTIONS:
Procedure: Epidural steroid with local anesthetic injection — Epidural steroid injectate will be 2cc of 1% lidocaine followed by 1-3 cc of 40 mg/cc Kenalog (i.e. 40-120 mg Kenalog) or an equivalent steroid medication (depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg) in an opaque syringe.
  Arms: Epidural Steroid injection
Procedure: Epidural local anesthetic injection — Epidural injectate will be 2cc of .25-1% lidocaine followed by 1-3cc of 1% lidocaine in an opaque syringe.
  Arms: Epidural local anesthetic injection
Drug: Epidural steroid injection — Epidural steroid injectate will be 2cc of .25 - 1% lidocaine followed by 1-3 cc of 40 mg/cc Kenalog (i.e. 40-120 mg Kenalog) or an equivalent steroid medication (depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg) in an opaque syringe.
  Other Names: Kenalog, depo-medrol, betamethasone or dexamethasone
  Arms: Epidural Steroid injection
Drug: Epidural local anesthetic injection — Epidural injectate will be 2cc of .25-1% lidocaine followed by 1-3cc of 1% lidocaine in an opaque syringe.
  Other Names: lidocaine
  Arms: Epidural local anesthetic injection

SUMMARY:
The broad, long-term objective of this research protocol is to improve the quality of life for patients suffering from lumbar spinal stenosis. This objective will be met by examining the safety and clinical efficacy of epidural steroid injections for treatment of pain associated with lumbar spinal stenosis. This prospective, randomized, double-blind controlled trial (RCT) will test the hypothesis that the effectiveness of epidural steroid injections (ESI) plus local anesthetic (LA) is greater than epidural injections of LA alone in older adults with lumbar spinal stenosis.

DETAILED DESCRIPTION:
Lumbar spinal stenosis is one of the most common causes of low back pain in the elderly and can lead to significant disability. The symptoms of spinal stenosis range from low back pain to neurogenic claudication with lower extremity pain, weakness and/or sensory changes related to activities. As spinal stenosis can affect the central canal as well as the lateral recesses and intervertebral foramen variably, symptoms can involve single or multiple myotomes and dermatomes. Since the causes of spinal stenosis are most frequently degenerative changes, the symptoms of spinal stenosis often, but not always, worsen over time. Despite the prevalence of spinal stenosis, treatment of spinal stenosis remains somewhat controversial. Common treatments include conservative measures such as non-steroidal anti-inflammatories (NSAIDS), activity modification and physical therapy as well as more invasive treatments such as epidural steroid injections and surgery. Although surgery has been demonstrated to provide some benefit to many individuals with spinal stenosis, ESI are being used with increasing frequency as a less invasive, potentially more cost effective and safer treatment for spinal stenosis. However, there is a lack of data to demonstrate the effectiveness and safety of epidural steroid injections for spinal stenosis, particularly in the older adults.

Because of the compelling need for effective therapy for patients suffering from spinal stenosis and because epidural steroid injections are rapidly becoming standard of care for treating these patients - even in the absence of compelling clinical evidence - we are conducting a randomized, controlled trial in order to test the hypothesis that lumbar epidural steroid injections improve functional status and pain associated with spinal stenosis. The main objective of the study is to conduct a blinded, randomized controlled trial (RCT) in elderly patients with spinal stenosis to test if the effectiveness of epidural steroid injections (ESI) plus local anesthetic (LA) is greater than LA alone.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the low back, buttock, and/or lower extremity (pain NRS>=5) with standing, walking and/or spinal extension (buttock/leg>back pain).
2. Modified Roland-Morris score of at least 7.
3. Mild-severe lumbar central canal spinal stenosis (Boden et al. criteria18) identified by MRI or CT scan.
4. Lower extremity symptoms consistent with neurogenic claudication.
5. Must be able to read English and complete the assessment instruments.
6. Age 50 or older.

Exclusion Criteria:

1. Cognitive impairment that renders the patient unable to give informed consent or provide accurate data.
2. Clinical co-morbidities that could interfere with the collection of data concerning pain and function.

   Known dx of fibromyalgia, chronic widespread pain, amputees, parkinsons, head injury, dementia, stroke, other neurologic conditions Collect date about cervical spinal stenosis, painful peripheral neuropathy, EMGs
3. Severe vascular, pulmonary or coronary artery disease that limits ambulation including recent myocardial infarction (within 6 months).
4. Spinal instability requiring surgical fusion.
5. Severe osteoporosis as defined by multiple compression fractures or a fracture at the same level as the stenosis.
6. Metastatic cancer.
7. Excessive alcohol consumption or evidence of non-prescribed or illegal drug use.
8. Possible pregnancy or other reason that precludes the use of fluoroscopy.
9. Concordant pain with internal rotation of the hip (or known hip joint pathology).
10. Active local or systemic infection.
11. Abnormal coagulation.
12. Allergy to local anesthetic, steroid or contrast.
13. Previous lumbar spine surgery.
14. Epidural steroid injection within previous 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janna L Friedly, MD, Principal Investigator — University of Washington
Locations (10):
- United States (10):
  - Kaiser Permanente Northern California, Redwood City, California
  - Kaiser Permanente Northern California, Roseville, California
  - University of Colorado, Denver, Colorado
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - Dallas VA Medical Center, Dallas, Texas
  - Virginia Spine Research Institute, Richmond, Virginia
  - Harborview Medical Center, University of Washington, Seattle, Washington

REFERENCES:
- [Background] Friedly JL, Bresnahan BW, Comstock B, Turner JA, Deyo RA, Sullivan SD, Heagerty P, Bauer Z, Nedeljkovic SS, Avins AL, Nerenz D, Jarvik JG. Study protocol- Lumbar Epidural steroid injections for Spinal Stenosis (LESS): a double-blind randomized controlled trial of epidural steroid injections for lumbar spinal stenosis among older adults. BMC Musculoskelet Disord. 2012 Mar 29;13:48. doi: 10.1186/1471-2474-13-48. PMID 22458343
- [Result] Turner JA, Comstock BA, Standaert CJ, Heagerty PJ, Jarvik JG, Deyo RA, Wasan AD, Nedeljkovic SS, Friedly JL. Can patient characteristics predict benefit from epidural corticosteroid injections for lumbar spinal stenosis symptoms? Spine J. 2015 Nov 1;15(11):2319-31. doi: 10.1016/j.spinee.2015.06.050. Epub 2015 Jun 19. PMID 26096484
- [Result] Suri P, Pashova H, Heagerty PJ, Jarvik JG, Turner JA, Comstock BA, Bauer Z, Annaswamy TM, Nedeljkovic SS, Wasan AD, Friedly JL. Short-term improvements in disability mediate patient satisfaction after epidural corticosteroid injections for symptomatic lumbar spinal stenosis. Spine (Phila Pa 1976). 2015 Sep 1;40(17):1363-70. doi: 10.1097/BRS.0000000000001000. PMID 26010037
- [Result] Friedly JL, Comstock BA, Turner JA, Heagerty PJ, Deyo RA, Sullivan SD, Bauer Z, Bresnahan BW, Avins AL, Nedeljkovic SS, Nerenz DR, Standaert C, Kessler L, Akuthota V, Annaswamy T, Chen A, Diehn F, Firtch W, Gerges FJ, Gilligan C, Goldberg H, Kennedy DJ, Mandel S, Tyburski M, Sanders W, Sibell D, Smuck M, Wasan A, Won L, Jarvik JG. A randomized trial of epidural glucocorticoid injections for spinal stenosis. N Engl J Med. 2014 Jul 3;371(1):11-21. doi: 10.1056/NEJMoa1313265. PMID 24988555
- [Derived] Friedly JL, Comstock BA, Turner JA, Heagerty PJ, Deyo RA, Bauer Z, Avins AL, Nedeljkovic SS, Nerenz DR, Shi XR, Annaswamy T, Standaert CJ, Smuck M, Kennedy DJ, Akuthota V, Sibell D, Wasan AD, Diehn F, Suri P, Rundell SD, Kessler L, Chen AS, Jarvik JG. Long-Term Effects of Repeated Injections of Local Anesthetic With or Without Corticosteroid for Lumbar Spinal Stenosis: A Randomized Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1499-1507.e2. doi: 10.1016/j.apmr.2017.02.029. Epub 2017 Apr 8. PMID 28396242

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Steroid Injection: Intervention: Epidural steroid with local anesthetic injection
  2cc of .25 - 1% lidocaine and glucocorticoid (Kenalog 40-120 mg, depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg)in an opaque syringe.
  Epidural steroid with local anesthetic injection: Epidural steroid injectate will be 2cc of 1% lidocaine followed by 1-3 cc of 40 mg/cc Kenalog (i.e. 40-120 mg Kenalog) or an equivalent steroid medication (depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg) in an opaque syringe.
  Epidural steroid injection: Epidural steroid injectate will be 2cc of .25 - 1% lidocaine followed by 1-3 cc of 40 mg/cc Kenalog (i.e. 40-120 mg Kenalog) or an equivalent steroid medication (depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg) in an opaque syringe.
Period: Overall Study
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection
Started | 200 | 200
Completed | 153 | 150
Not Completed | 47 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.8) | 68.1 (10.2) | 68 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 104 | 221
  Male | 83 | 96 | 179

OUTCOME MEASURES:

1. Primary Outcome: Roland Morris
Description: The primary outcome measure will be back specific functional status, measured by the Roland Scale at 6 weeks. The RDQ is a back pain specific functional status questionnaire adapted from the Sickness Impact Profile (SIP). The RDQ consists of 24 yes/no items, which represent common dysfunctions in daily activities experienced by subjects with low back pain. A single unweighted score is derived by summing the 24 items, with higher scores indicating worse function with 0 (no disability) to 24 (maximum disability). Our primary analysis will be a simple 2-group comparison of the mean Roland score as an evaluation of the short-term efficacy of epidural steroid injection.
Time Frame: 6 weeks
Population: 6 week follow up rate was 97% (n=193/200, n=193/200).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection
Number analyzed (Participants) | 193 | 193
units on a scale | 11.8 (6.3) | 12.5 (6.4)

2. Secondary Outcome: Pain Numeric Rating Scale
Description: Leg Pain NRS is a second primary outcome at 6 weeks We measured leg pain using a 0-10 pain NRS (0=no pain and 10=worst pain imaginable) assessing average pain over the past week.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection
Number analyzed (Participants) | 193 | 193
units on a scale | 4.4 (2.9) | 4.6 (2.9)

3. Secondary Outcome: Roland Morris Disability Questionnaire (RDQ)
Description: The RDQ is a back pain specific functional status questionnaire adapted from the Sickness Impact Profile (SIP). The RDQ consists of 24 yes/no items, which represent common dysfunctions in daily activities experienced by subjects with low back pain. A single unweighted score is derived by summing the 24 items, with higher scores indicating worse function with 0 (no disability) to 24 (maximum disability). Our primary analysis will be a simple 2-group comparison of the mean Roland score as an evaluation of the short-term efficacy of epidural steroid injection.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Epidural Steroid Injection: Intervention: Epidural steroid with local anesthetic injection
  2cc of .25 - 1% lidocaine and glucocorticoid (Kenalog 40-120 mg, depo-medrol 60-120 mg, betamethasone 6-12 mg or dexamethasone 8-10 mg)
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection
Number analyzed (Participants) | 180 | 174
units on a scale | 12.0 (6.5) | 11.5 (7.1)

4. Secondary Outcome: Leg Pain NRS
Description: Leg Pain NRS 0-10 scale
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection
Number analyzed (Participants) | 180 | 174
units on a scale | 4.7 (3.1) | 4.3 (3.1)

ADVERSE EVENTS:
Arm/Group | Epidural Steroid Injection | Epidural Local Anesthetic Injection
Serious Adverse Events (participants affected / at risk) | 5/200 | 4/200
Other Adverse Events (participants affected / at risk) | 43/200 | 31/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Steroid Injection (N=200) | Epidural Local Anesthetic Injection (N=200)
Hospitalization or Surgery (Surgical and medical procedures) | 5 (5) | 4 (4) — Any hospitalization or surgery was included as a serious adverse event. this included lumbar spine surgery for failure to improve symptoms or hospitalizations for any reason. None were deemed directly associated with the interventions.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Steroid Injection (N=200) | Epidural Local Anesthetic Injection (N=200)
Dural puncture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Dural puncture at time of procedure
All other self reported adverse events (General disorders) | 43 (57) | 31 (33) — Patients were asked an open-ended question about whether they experienced any adverse event or unexpected adverse event. Patients described the AE, but there were no consistent descriptions to clearly separate into rates for each type of AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days